CLINICAL TRIAL: NCT07052435
Title: Pressure (Fractional Flow Reserve) and Flow (Vascular Flow Reserve) Measurements During Peripheral Arterial Interventions
Acronym: FLOW-PAD
Status: Recruiting | Type: Observational
Sponsor: Dr. Konstantinos Katsanos (Other)
Collaborators: Medlytic Labs (Unknown); Attikon Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr. Konstantinos Katsanos, Professor, University Hospital of Patras
Organization: University Hospital of Patras (Other)
Other Study IDs: 422
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia (CLI)
Keywords: fractional flow reserve; coronary flow reserve; vascular flow reserve
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAD: Infrainguinal arterial occlusive disease presenting with intermittent claudication or critical limb ischemia

SUMMARY:
Fractional Flow Reserve (FFR) and Coronary Flow Reserve (CFR) have been originally developed for physiological assessment of coronary artery disease and may hold potential in the management of Peripheral Arterial Disease (PAD) as well. By adapting pressure and flow measurements for the peripheral arteries, clinicians could objectively evaluate stenosis severity, guiding treatment decisions and optimizing outcomes. The aim of this study is to evaluate the diagnostic performance of FFR and vascular Flow Reserve (VFR, aka CFR) for detection of functionally significant peripheral arterial disease and to derive appropriate cut-off values for the prediction of successful immediate and long-term clinical outcomes.

DETAILED DESCRIPTION:
Understanding Fractional Flow Reserve (FFR)

When it comes to diagnosing and managing coronary artery disease (CAD), medical advancements have introduced various tools and techniques to provide accurate assessments. One such critical method is Fractional Flow Reserve (FFR), a groundbreaking approach that aids physicians in making informed decisions regarding the necessity of coronary interventions.

What is Fractional Flow Reserve (FFR)?

Fractional Flow Reserve, commonly referred to as FFR, is a physiological index used to measure the severity of stenosis or narrowing in coronary arteries. It's a ratio of the maximum blood flow in a stenotic artery to the maximum blood flow if that artery if it were unobstructed. In simpler terms, FFR helps determine if a particular blockage in the coronary artery is significant enough to warrant intervention, such as angioplasty or stent placement.

How is FFR Measured?

FFR measurement is typically performed during a coronary angiogram, an imaging procedure that visualizes the blood vessels of the heart. A pressure-sensitive guidewire is threaded through the coronary arteries to reach the area of interest. By measuring the pressure before and after the stenosis, FFR is calculated as the ratio of distal (post-stenotic) pressure to proximal (pre-stenotic) pressure. An FFR value of 1 indicates no significant obstruction, while a value less than 0.80 is considered indicative of a hemodynamically significant stenosis that may benefit from intervention.

Significance in Clinical Decision-Making

The introduction of FFR has revolutionized the management of CAD. Prior to FFR, decisions about which stenoses to treat were often based solely on visual assessment during coronary angiography. However, studies have shown that visual assessments can sometimes be inaccurate, leading to unnecessary interventions. FFR provides objective physiological data that guides clinicians in identifying lesions that truly require treatment, thereby reducing the number of unnecessary procedures.

Applications and Advantages of Fractional Flow Reserve

Clinical Applications

1. Treatment Selection: FFR has become an essential tool in determining the necessity of revascularization procedures such as angioplasty and stenting. It helps clinicians differentiate between lesions that are causing significant blood flow restrictions and those that can be safely managed with medical therapy alone.
2. Risk Stratification: FFR aids in risk assessment by identifying high-risk lesions that are more likely to cause adverse cardiac events. This enables healthcare providers to prioritize interventions for patients at greater risk, improving patient outcomes.
3. Multi-Vessel Disease Management: In patients with multi-vessel coronary artery disease, FFR assists in deciding which vessel to treat first. By evaluating the functional significance of each stenosis, physicians can adopt a more tailored and effective treatment strategy.

Advantages of FFR

1. Evidence-Based Decision-Making: FFR provides objective physiological data, reducing subjectivity in treatment decisions. This evidence-based approach enhances patient care by ensuring that interventions are performed only when clinically necessary.
2. Cost-Efficiency: By avoiding unnecessary interventions, FFR helps optimize healthcare costs. Patients who do not require interventions based on FFR results can be managed conservatively, saving resources without compromising care quality.
3. Improved Patient Outcomes: As FFR assists in identifying lesions with the greatest impact on blood flow, interventions are more likely to be successful in restoring optimal blood flow. This translates to improved patient outcomes and quality of life.

Fractional Flow Reserve (FFR) has emerged as a game-changer in the field of cardiology, transforming how coronary artery disease is diagnosed and managed. By providing objective physiological data about the severity of stenosis, FFR enables clinicians to make informed decisions about treatment interventions. Its impact extends beyond reducing unnecessary procedures to enhancing patient outcomes, optimizing healthcare costs, and facilitating personalized treatment plans. As technology continues to evolve, FFR remains a cornerstone of modern cardiology, ensuring that patients receive the most effective and appropriate care for their coronary artery disease.

Exploring the Potential Use of FFR and CFR in Peripheral Arterial Disease (PAD)

While Fractional Flow Reserve (FFR) and Coronary Flow Reserve (CFR) have primarily found their applications in diagnosing and managing coronary artery disease (CAD), their potential utility could possibly extend beyond the realm of the heart. Peripheral Arterial Disease (PAD), a condition involving narrowed arteries outside of the heart, can also benefit from the insights provided by FFR and CFR. In this study, we will delve into how FFR and CFR could revolutionize the assessment and treatment of PAD.

Peripheral Arterial Disease (PAD) and Its Challenges

PAD is characterized by atherosclerotic plaque buildup in arteries supplying blood to the extremities, particularly the legs. This condition leads to reduced blood flow, which can cause pain, impaired wound healing, and even limb-threatening complications. Accurate assessment of the severity of arterial blockages and the evaluation of microvascular function are critical in managing PAD effectively.

Adapting FFR to Peripheral Arteries

While FFR is commonly used in coronary arteries, a very promising application could be its deployment in peripheral arteries. The principle remains the same: measuring pressure gradients across a stenosis to determine its functional significance. FFR can be adapted to assess stenosis severity in peripheral arteries, in an attempt helping clinicians decide whether interventions such as angioplasty or stenting are necessary.

Plausible Benefits in PAD Assessment

The application of FFR in PAD assessment may offer several benefits:

* Objective Assessment: FFR could provide objective physiological data, reducing subjectivity in determining which arterial stenoses are truly obstructive and require intervention.
* Guiding Treatment Decisions: By accurately identifying lesions that impact blood flow, FFR assists in guiding treatment decisions, ensuring that interventions are targeted and effective.
* Reducing Unnecessary Interventions: Like in CAD, FFR could help avoid unnecessary procedures in PAD, improving patient outcomes and conserving healthcare resources.

Leveraging CFR for Microvascular Assessment in PAD, Coronary Flow Reserve (CFR) in PAD - Microvascular Dysfunction in PAD

While CFR is commonly associated with coronary microvascular function, its application can be extended to assess microvascular function in peripheral arteries affected by PAD. Microvascular dysfunction plays a crucial role in PAD-related symptoms and complications, including poor wound healing and ischemic pain.

Evaluating Microvascular Function By assessing blood flow under both resting and stress conditions, clinicians can evaluate the ability of microvasculature to respond to increased demand.

Significance in PAD Management

CFR's role in assessing microvascular function can provide valuable insights:

* Early Detection of Dysfunction: Reduced CFR in peripheral arteries may indicate microvascular dysfunction before the onset of severe symptoms. Early detection allows for proactive management.
* Tailoring Treatment Strategies: Patients with PAD and microvascular dysfunction might require unique treatment approaches, such as medications targeting microcirculatory function, alongside interventions addressing larger arterial blockages.

Conclusion Fractional Flow Reserve (FFR) and Coronary Flow Reserve (CFR), originally developed for coronary artery assessment, hold tremendous potential in revolutionizing the management of Peripheral Arterial Disease (PAD). By adapting FFR for peripheral arteries, clinicians could objectively evaluate stenosis severity, guiding treatment decisions and optimizing outcomes. Leveraging CFR to assess microvascular function in peripheral arteries offers insights into early-stage dysfunction and aids in tailoring treatment strategies. As the medical field evolves, the integration of FFR and CFR into PAD management showcases the power of innovative techniques in enhancing patient care across diverse cardiovascular conditions.

Hypothesis and study design We hypothesized that the measurement of physiological indices FFR and CFR during peripheral angioplasty of the femoropopliteal segment may optimize procedural outcomes and improve long-term clinical results. This is a cohort study with some 100 patients suffering from PAD (both claudicants and patients with critical ischemia) to be recruited for FFR and CFR measurements before and after definitive endovascular intervention in parallel with standard angiographic control. CFR will be measured with an artificial intelligence computer model (Medlytic Labs) employing reduced-order navier Stokes equations and angiographic images validated against Doppler based velocity measurements at rest and hyperemia.

The aim of this study is to evaluate the diagnostic performance of FFR and peripheral Vascular Flow reserve (VFR, aka CFR) for detection of functionally significant peripheral arterial disease and to derive appropriate cut-off values for the prediction of successful immediate and long-term clinical outcomes. Patients will be observed long-term and we will keep records of any future TLF (target lesion failure), MACE (major adverse cardiovascular event) or MALE (major adverse limb event) during the whole follow-up period. The follow-up time will be 24 months and events will be captured and analyzed with time-to-event methods.

The primary outcomes of interest in this study will include:

1. the treated target lesion failure (TLF) as defined below.
2. any MACE event during the follow-up observation period as defined below.
3. any MALE event during the follow-up observation period as defined below. FFR and CFR will be recorded with the application of guideline-recommended standard of care methods in line with coronary practice. We will analyze the diagnostic performance of FFR and CFR with standard receiver-operating characteristic curves using Rutherford stage symptoms combined with ankle-brachial index as a reference test. In addition, we will regress above endpoints with appropriate Cox models to derive relevant predictors of long-term clinical results.

TLF (Target lesion failure) is defined as the composite of clinically driven TLR (Target lesion revascularization), acute limb ischemia or vascular amputation related to the target vessel. Target lesion is the segment where intervention was performed, and the length of the target lesion is inclusive of the arterial segment treated. Target vessel is the major native femoropopliteal axis or bypass graft containing the target lesion. If it cannot be determined with certainty whether an acute limb ischemia or vascular amputation is related to the target vessel, and at the same time if no other specific reasons can be given, it will be considered as a case of MALE.

MALE (major adverse limb events) is defined as acute or chronic limb ischemia, including major vascular amputation.

Acute limb ischemia was defined as limb threatening ischemia that was confirmed by using limb hemodynamic parameters or imaging and led to an acute vascular intervention (pharmacological [heparin, thrombolysis], peripheral artery surgery/reconstruction, peripheral angioplasty/stent, or amputation) within 30 days of onset of symptoms.

Chronic limb ischemia was defined as continuing ischemic limb, foot, or digit pain leading to hospitalization and intervention and not meeting the definition of acute limb ischemia.

Patients with Fontaine classification III or IV at baseline, who had a peripheral vascular intervention.

Major vascular amputation was defined as an amputation due to a vascular event above the forefoot.

Peripheral vascular interventions were defined as interventions (including peripheral angioplasty, vascular surgery, or amputation) not meeting the definition for acute limb ischemia or chronic limb ischemia.

MACE (major adverse cardiovascular events) is defined as cardiovascular death, non-fatal myocardial infraction, non-fatal stroke and percutaneous or surgical coronary revascularization procedures.

Cardiovascular Death: This refers to death caused by a cardiovascular event, such as a heart attack, heart failure, arrhythmia, or other heart-related causes.

Non-Fatal Myocardial Infarction: An MI occurs when there is a blockage of blood flow to a portion of the heart muscle, leading to ischemia.

Non-Fatal Stroke: A stroke happens when blood flow to a part of the brain is disrupted, causing brain cells to be damaged or die.

Coronary revascularization procedures (e.g., angioplasty or coronary artery bypass graft surgery).

ELIGIBILITY:
Inclusion Criteria:

Symtpomatic peripheral arterial disease. Intermittent claudication or critical limb ischemia. Documented steno-occlusive disease of the femoropopliteal segment by imaging. Provision of informed consent form.

Exclusion Criteria:

Aortoiliac occlusive disease. Acute limb ischemia. Aneurysmal infrainguinal disease. General contra-indications to percutaneous ballon angioplasty and/or other endovascular procedures like dementia or bleeding diathesis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering with symptoms of peripheral arterial disease (intermittent claudication or critical limb ischemia) and opting for endovascular treatment of infrainguinal arterial occlusive disease documented by Duplex ultrasound or cross-sectional imaging.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
TLF (Target lesion failure) | 24 months
  TLF (Target lesion failure) is defined as the composite of clinically driven TLR (Target lesion revascularization), acute limb ischemia or vascular amputation related to the target vessel. Target lesion is the segment where intervention was performed, and the length of the target lesion is inclusive of the arterial segment treated. Target vessel is the major native femoropopliteal axis or bypass graft containing the target lesion.

SECONDARY OUTCOMES:
MALE (major adverse limb events) | 24 months
  MALE (major adverse limb events) is defined as acute or chronic limb ischemia, including major vascular amputation.
  Acute limb ischemia was defined as limb threatening ischemia that was confirmed by using limb hemodynamic parameters or imaging and led to an acute vascular intervention (pharmacological [heparin, thrombolysis], peripheral artery surgery/reconstruction, peripheral angioplasty/stent, or amputation) within 30 days of onset of symptoms.
  Chronic limb ischemia was defined as continuing ischemic limb, foot, or digit pain leading to hospitalization and intervention and not meeting the definition of acute limb ischemia.
  Patients with Fontaine classification III or IV at baseline, who had a peripheral vascular intervention.
  Major vascular amputation was defined as an amputation due to a vascular event above the forefoot.
  Peripheral vascular interventions were defined as interventions (including peripheral angioplasty, vascular surgery, or amputation) not meeting the definition
MACE (major adverse cardiovascular events) | 24 months
  MACE (major adverse cardiovascular events) is defined as cardiovascular death, non-fatal myocardial infraction, non-fatal stroke and percutaneous or surgical coronary revascularization procedures.
  Cardiovascular Death: This refers to death caused by a cardiovascular event, such as a heart attack, heart failure, arrhythmia, or other heart-related causes.
  Non-Fatal Myocardial Infarction: An MI occurs when there is a blockage of blood flow to a portion of the heart muscle, leading to ischemia.
  Non-Fatal Stroke: A stroke happens when blood flow to a part of the brain is disrupted, causing brain cells to be damaged or die.
  Coronary revascularization procedures (e.g., angioplasty or coronary artery bypass graft surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: No